CLINICAL TRIAL: NCT03351075
Title: The Effectiveness of a Modern Educational Intervention for Pain-related Disability After Breast Cancer Surgery: Randomized Controlled Trial
Brief Title: Effectiveness of a Modern Educational Intervention in Breast Cancer Patients
Acronym: EduCan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: s60702
Record Dates: First submitted 2017-10-04; First posted 2017-11-22 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2022-05

CONDITIONS: Breast Neoplasm; Pain
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Standard physical therapy program + Modern educational program
  Interventions: Other: Standard physical therapy program; Other: Modern educational program
- Control group (Active Comparator): Standard physical therapy program + Traditional biomedical educational program
  Interventions: Other: Standard physical therapy program; Other: Traditional biomedical educational program

INTERVENTIONS:
Other: Standard physical therapy program — Mobilisations, stretching, scar tissue treatment and exercises
  * Start immediately after surgery, sessions are individual and take 30 minutes
  * Intensive phase (4 months): 1-2x/week
  * Maintenance phase (8 months, 3 sessions): 6, 8 and 12 months post-surgery
Other: Modern educational program — This modern neuroscience educational approach is suited to explain more complex issues associated with pain such as the involvement of peripheral and central mechanisms, neuroplasticity and pain behaviour.
  * Sessions are individual and take 30 minutes, in addition to the standard physical therapy sessions
  * 3 sessions during week 1-2, 3 booster sessions at 6, 8 and 12 months post-surgery
  Arms: Intervention group
Other: Traditional biomedical educational program — Traditional educational interventions are applied according to the biomedical model. This means that the patient's pain experience is explained from a tissue (injured versus healthy tissue) and biomechanics perspective
  * Sessions are individual and take 30 minutes, in addition to the standard physical therapy sessions
  * 3 sessions during week 1-2, 3 booster sessions at 6, 8 and 12 months post-surgery
  Arms: Control group

SUMMARY:
In addition to fatigue, pain is the most frequent and persistent symptom following breast cancer and breast cancer treatment. Despite the effectiveness of different physical therapy modalities, such as manual techniques, passive mobilizations and exercises, many patients still experience pain and subsequent difficulties in daily functioning at short and long term. Past decades, the awareness on the important role of educational interventions in the management of pain in general has increased. Educational interventions aim at explaining and improving the knowledge, control and attitude of the patient regarding his/her pain complaint. However, these educational interventions are often restricted to more biomedical pain management instructions and general advice on physical activity and analgesics (= traditional biomedical education). Only recently, increased knowledge on pain mechanisms led to a more modern educational approach. This modern approach is suited to explain more complex issues associated with pain and takes into account many more factors related to pain. To our knowledge, only one controlled trial investigated the effectiveness of a modern educational intervention in the early stage of breast cancer treatment. The results were very promising for shoulder function. However, only short-term effects were examined, no randomization was performed and no pain-related and socio-economic outcomes were evaluated. Therefore, the aim of the proposed project is to investigate the effectiveness of a similar modern educational program, in addition to standard physical therapy care, in the early treatment phase of breast cancer in comparison with traditional biomedical education. A randomized controlled trial will be performed with a long-term follow up period. The primary outcome parameter is pain-related disability. Secondary outcomes are different dimensions of pain, physical and mental functioning, return to work and health-care related costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary breast cancer
* Unilateral surgery including, either:

Axillary lymph node dissection and mastectomy/breast -conserving/reconstructive surgery OR Sentinel Node Biopsy and mastectomy/reconstructive surgery

Exclusion Criteria:

* Active metastasis
* Cannot participate during the entire study period

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lore Dams, Dra, Principal Investigator — University of Leuven; Elien Van der Gucht, Dra, Principal Investigator — University of Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Background] De Groef A, Devoogdt N, Van der Gucht E, Dams L, Bernar K, Godderis L, Morlion B, Moloney N, Smeets A, Van Wilgen P, Meeus M. EduCan trial: study protocol for a randomised controlled trial on the effectiveness of pain neuroscience education after breast cancer surgery on pain, physical, emotional and work-related functioning. BMJ Open. 2019 Jan 4;9(1):e025742. doi: 10.1136/bmjopen-2018-025742. PMID 30612114
- [Result] Dams L, Van der Gucht E, Devoogdt N, Smeets A, Bernar K, Morlion B, Godderis L, Haenen V, De Vrieze T, Fieuws S, Moloney N, Van Wilgen P, Meeus M, De Groef A. Effect of pain neuroscience education after breast cancer surgery on pain, physical, and emotional functioning: a double-blinded randomized controlled trial (EduCan trial). Pain. 2023 Jul 1;164(7):1489-1501. doi: 10.1097/j.pain.0000000000002838. Epub 2022 Dec 8. PMID 36637138
- [Result] Dams L, Van der Gucht E, Haenen V, Devoogdt N, Smeets A, Bernar K, Morlion B, Moloney N, Fieuws S, De Groef A, Meeus M. Effectiveness of pain neuroscience education on somatosensory functioning after surgery for breast cancer: A double-blinded randomized controlled trial. Anat Rec (Hoboken). 2024 Feb;307(2):248-272. doi: 10.1002/ar.25127. Epub 2023 Jan 3. PMID 36594663
- [Result] De Groef A, Van der Gucht E, Devoogdt N, Smeets A, Bernar K, Morlion B, Godderis L, De Vrieze T, Fieuws S, Meeus M, Dams L. Returning to Work After Breast Cancer Surgery: A Randomised Controlled Trial on the Effect of Pain Neuroscience Education. J Occup Rehabil. 2023 Dec;33(4):757-765. doi: 10.1007/s10926-023-10103-9. Epub 2023 May 12. PMID 37171771
- [Derived] Amber G, Lore D, Elien VG, Jan S, Michel M, An G, Mira M. From breast cancer diagnosis to survivorship: Analyzing perioperative biopsychosocial phenotypes and their relationship to pain on long term. J Pain. 2025 Jan;26:104709. doi: 10.1016/j.jpain.2024.104709. Epub 2024 Oct 16. PMID 39419367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the Multidisciplinary Breast Center of the University Hospitals Leuven campus Gasthuisberg (Belgium) between November 2017 and March 2020.
Pre-assignment Details: In total, 493 women were eligible, of which 184 were included in the study.
Groups:
- Intervention Group: Standard physical therapy program + Modern educational program
  Standard physical therapy program: Mobilisations, stretching, scar tissue treatment and exercises
  * Start immediately after surgery, sessions are individual and take 30 minutes
  * Intensive phase (4 months): 1-2x/week
  * Maintenance phase (8 months, 3 sessions): 6, 8 and 12 months post-surgery
  Modern educational program: This modern neuroscience educational approach is suited to explain more complex issues associated with pain such as the involvement of peripheral and central mechanisms, neuroplasticity and pain behaviour.
  * Sessions are individual and take 30 minutes, in addition to the standard physical therapy sessions
  * 3 sessions during week 1-2, 3 booster sessions at 6, 8 and 12 months post-surgery
- Control Group: Standard physical therapy program + Traditional biomedical educational program
  Standard physical therapy program: Mobilisations, stretching, scar tissue treatment and exercises
  * Start immediately after surgery, sessions are individual and take 30 minutes
  * Intensive phase (4 months): 1-2x/week
  * Maintenance phase (8 months, 3 sessions): 6, 8 and 12 months post-surgery
  Traditional biomedical educational program: Traditional educational interventions are applied according to the biomedical model. This means that the patient's pain experience is explained from a tissue (injured versus healthy tissue) and biomechanics perspective
  * Sessions are individual and take 30 minutes, in addition to the standard physical therapy sessions
  * 3 sessions during week 1-2, 3 booster sessions at 6, 8 and 12 months post-surgery
Period: Intensive Treatment Phase (4 mo FU)
Arm/Group | Intervention Group | Control Group
Started | 92 | 92
Completed | 86 | 87
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Death | 0 | 1
Period: Maintenance Treatment Phase (12 mo FU)
Arm/Group | Intervention Group | Control Group
Started | 86 | 87
Completed | 85 | 87
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: End of Trial (18 mo FU)
Arm/Group | Intervention Group | Control Group
Started | 85 | 87
Completed | 84 | 86
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 76 | 150
  >=65 years | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.5) | 55.2 (11.4) | 55.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 92 | 184
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 92 | 92 | 184
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (4.3) | 25.9 (5.9) | 25.6 (5.2)
Educational Level [Number; unit: participants] — Population: Assessed retrospectively at 4 months after surgery, so only calculated from data available at 4 months postoperatively. Missing data is present.
  participants
    Primary education or no diploma: number analyzed (Participants) | 86 | 87 | 173
    Primary education or no diploma | 3 | 3 | 6
    Lower secondary education: number analyzed (Participants) | 86 | 87 | 173
    Lower secondary education | 5 | 5 | 10
    Upper secondary education: number analyzed (Participants) | 86 | 87 | 173
    Upper secondary education | 23 | 28 | 51
    Higher education: professional bachelor: number analyzed (Participants) | 86 | 87 | 173
    Higher education: professional bachelor | 30 | 32 | 62
    Higher education: academic bachelor or master: number analyzed (Participants) | 86 | 87 | 173
    Higher education: academic bachelor or master | 25 | 19 | 44
Surgery at dominant side [Number; unit: participants]
  Surgery at dominant side (yes) | 44 | 41 | 85
  Surgery at dominant side (no) | 48 | 51 | 99
Type of surgery [Number; unit: participants] — ALND: axillary lymph node dissection, BCS: breast conserving surgery, ME=mastectomy, SLNB=Sentinel Lymph Node Biopsy
  participants
    BCS+ALND | 4 | 9 | 13
    1ME+SLNB | 41 | 43 | 84
    ME+ALND | 47 | 40 | 87
Radiotherapy [Number; unit: participants] | 74 | 66 | 140
Hormone therapy [Number; unit: participants] | 69 | 68 | 137
Chemotherapy [Number; unit: participants] | 63 | 55 | 118

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Change in Pain-related Disability
Description: Measured with Pain Disability Index, an instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. Scores between 0 and 70. The higher the score the greater the person's disability due to pain.
Time Frame: Change between baseline and one year follow-up assessment
Population: Using likelihood-based estimation, subjects with a missing at one or more timepoints were still included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 82 | 84
score on a scale | 4.22 [1.40 to 7.03] | 5.53 [2.74 to 8.32]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; The sample size was based on comparing the changes for the primary outcome measure (PDI-DLV) at 12 months after surgery. The calculation was based on comparing the values at 12 months. Assuming a coefficient of variation (CV) equal to 0.5, 87 participants per group were needed based on a two-sample pooled t-test of a mean ratio with lognormal data and α=0.05 to detect with 80% power a difference of 20% in PDI. To anticipate a drop-out ratio of 5%, a total of 184 subjects were needed; Test type: Superiority; p = 0.5163, Multivariate linear model — No corrections for multiple testing were performed; A multivariate linear model for longitudinal measures with an unstructured covariance matrix was applied for each continuous outcome; Mean Difference (Net) = -1.31, 95% CI 2-sided [-5.28 to 2.65]

2. Secondary Outcome: Self-reported Pain-related Disability
Description: as for outcome 1
Time Frame: Postoperatively after 4 months of intensive treatment and at 1,5 years (after follow-up)
Population: Available data differed between timepoints
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Change from baseline to 4 months: number analyzed (Participants) | 88 | 89
  Change from baseline to 4 months | 3.70 [1.37 to 6.04] | 4.67 [2.35 to 6.99]
  Change from baseline to 1.5 years: number analyzed (Participants) | 83 | 86
  Change from baseline to 1.5 years | 3.13 [0.59 to 5.67] | 4.19 [1.68 to 6.70]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain-related disability from baseline to 4 months; Test type: Superiority; p = 0.5655, multivariate linear model — No corrections for multiple testing were performed; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.97, 95% CI 2-sided [-4.26 to 2.33]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain-related disability from baseline to 1.5 years; Test type: Superiority; p = 0.5592, multivariate linear model — P<.05 was considered significant. No corrections for multiple testing were performed; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.07, 95% CI 2-sided [-4.64 to 2.51]

3. Secondary Outcome: Self-reported Pain-intensity
Description: Measured with Visual Analogue Scale (0-100), lower scores indicate a better outcome.
Time Frame: Postoperatively after 4 months of intensive treatment, at 1 year (after maintenance treatment) and at 1,5 years (after follow-up)
Population: Available data differed between timepoints.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 88 | 89
  Mean change from baseline to 4 months | 7.26 [1.87 to 12.65] | 9.49 [4.14 to 14.85]
  Mean change from baseline to 12 months: number analyzed (Participants) | 81 | 84
  Mean change from baseline to 12 months | 6.31 [1.06 to 11.57] | 10.61 [5.43 to 15.79]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 83 | 86
  Mean change from baseline to 1.5 years | 3.91 [-1.70 to 9.52] | 8.71 [3.17 to 14.24]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain intensity from baseline to 4 months; Test type: Superiority; p = 0.5630, Multivariate linear model — No corrections for multiple testing were performed; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.23, 95% CI 2-sided [-9.84 to 5.37]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain intensity from baseline to 12 months; Test type: Superiority; p = 0.2524, Multivariate linear model — No corrections for multiple testing were performed; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.30, 95% CI 2-sided [-11.68 to 3.09]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain intensity from baseline to 1.5 years; Test type: Superiority; p = 0.2315, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.80, 95% CI 2-sided [-12.69 to 3.09]

4. Secondary Outcome: Self-reported Central Sensitization Symptoms
Description: Measured with the Central Sensitization Inventory (0-100). The Central Sensitization Inventory (CSI) includes 25 items about symptoms related to altered central somatosensory functioning, scored on a five-point Likert scale from 0 (never) to 4 (always). Scores range from 0-100 and a higher score represents greater symptomatology associated with altered central somatosensory processing.
Time Frame: as for outcome 3
Population: Available data differed on timepoints
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 80 | 86
  Mean change from baseline to 4 months | 3.61 [1.56 to 5.66] | 3.43 [1.15 to 5.14]
  Mean change from baseline to 1 year: number analyzed (Participants) | 82 | 81
  Mean change from baseline to 1 year | 2.14 [0.13 to 4.16] | 2.39 [0.40 to 4.38]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 79 | 83
  Mean change from baseline to 1.5 years | 3.15 [1.09 to 5.20] | 3.43 [1.15 to 5.14]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported central sensitisation symptoms from baseline to 4 months; Test type: Superiority; p = 0.7494, Multivariate linear model — No corrections for multiple testing were performed; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.47, 95% CI 2-sided [-2.39 to 3.32]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; The difference in change in self-reported central sensitisation symptoms from baseline to 12 months; Test type: Superiority; p = 0.8617, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.25, 95% CI 2-sided [-3.09 to 2.58]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported central sensitisation symptoms from baseline to 1.5 years; Test type: Superiority; p = 0.8454, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.29, 95% CI 2-sided [-3.16 to 2.59]

5. Secondary Outcome: Altered Somatosensory Functions (Touch)
Description: Mechanical detection sensitivity (mN) measured with Von Frey monofilaments at the arm at the affected side. A series of stimulus intensities are given and the stimulus intensity (mN) that is first identified is recorded (min-max 8 mN-512 mN). A lower value indicates a higher sensitivity to mechanical sensitivity.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: mN
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
mN
  Mean change from baseline to 4 months: number analyzed (Participants) | 83 | 92
  Mean change from baseline to 4 months | 2.37 [1.53 to 3.67] | 1.76 [1.13 to 2.72]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 69
  Mean change from baseline to 1 year | 1.68 [1.06 to 2.67] | 1.95 [1.22 to 3.09]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 80
  Mean change from baseline to 1.5 years | 2.35 [1.48 to 3.74] | 1.87 [1.18 to 2.95]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in mechanical detection sensitivity at the arm from baseline to 4 months; Test type: Superiority; p = 0.3463, multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.35, 95% CI 2-sided [0.72 to 2.51]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in mechanical detection sensitivity at the arm from baseline to 1 year; Test type: Superiority; p = 0.6613, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.86, 95% CI 2-sided [0.451 to 1.66]
Statistical Analysis 3: Comparison: Intervention Group; Difference in change in mechanical detection sensitivity at the arm from baseline to 1.5 years; Test type: Superiority; p = 0.4908, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.26, 95% CI 2-sided [0.65 to 2.42]

6. Secondary Outcome: Altered Somatosensory Functions (Temperature-warmth)
Description: Thermal detection sensitivity (degrees Celsius) for warmth at the arm at the affected side measured with computerized thermotests. Temperature when a change from a thermoneutral state to a distinct warm is recorded. A lower value indicates a higher sentivity to temperature.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: degrees celcius
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
degrees celcius
  Mean change from baseline to 4 months: number analyzed (Participants) | 83 | 82
  Mean change from baseline to 4 months | 3.54 [2.51 to 4.57] | 3.32 [2.28 to 4.36]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 68
  Mean change from baseline to 1 year | 2.67 [1.60 to 3.74] | 2.38 [1.30 to 3.45]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 80
  Mean change from baseline to 1.5 years | 2.74 [1.74 to 3.74] | 2.72 [1.74 to 3.70]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in warmth detection sensitivity from baseline to 4 months; Test type: Superiority; p = 0.7708, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.22, 95% CI 2-sided [-1.25 to 1.69]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in warmth detection sensitivity from baseline to 1 year; Test type: Superiority; p = 0.7060, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.29, 95% CI 2-sided [-1.23 to 1.81]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in warmth detection sensitivity from baseline to 1.5 years; Test type: Superiority; p = 0.9806, Multivariate linear model; Mean Difference (Net) = 0.02, 95% CI 2-sided [-1.38 to 1.42]

7. Secondary Outcome: Endogenous Pain Facilitation Assessed by a Temporal Summation Paradigm (0-10)
Description: Measured with repetitive pinprick stimuli (using Von Frey Monofilament of 256 mN) at the pectoral region of the affected side. Pain rating after a single stimulation and after 30s of stimulation is recorded. The outcome of interest is the pain rating after 30s stimulation - pain rating single stimulation on a Numeric Rating Scale (0-10) with lower scores meaning less endogenous pain facilitation.
Time Frame: as for outcome 3
Population: Available data differs per timepoints
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 83 | 82
  Mean change from baseline to 4 months | 0.95 [0.48 to 1.41] | 0.21 [-0.26 to 0.68]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 68
  Mean change from baseline to 1 year | 0.24 [-021 to 0.69] | 0.15 [-0.30 to 0.60]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 80
  Mean change from baseline to 1.5 years | 0.48 [-0.02 to 0.97] | 0.17 [-0.32 to 0.65]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in wind-up from baseline to 4 months; Test type: Superiority; p = 0.0284, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.74, 95% CI 2-sided [0.08 to 1.40]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in wind-up from baseline to 1 year; Test type: Superiority; p = 0.7776, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.55 to 0.73]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in wind-up from baseline to 1.5 years; Test type: Superiority; p = 0.3829, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.39 to 1.01]

8. Secondary Outcome: Endogenous Pain Inhibition Assessed by a Conditioned Pain Modulation Paradigm (0-10)
Description: Conditioned Pain Modulation Measured with TSA-II NeuroSensory Analyzer from Medoc. Parallel heat design is used with
  1. Test stimulus (45s): Individually determined test stimulus (temperature with a Numeric Rating Scale score of at least 4 out of 10) applied alone. Pain rating (Numeric Rating Scale 0-10) at 10s, 20s, 30s and 40s of stimulation.
  2. Break (120s)
  3. Conditioning stimulus (temperature of test stimulus + 0.5°C) (65s) + test stimulus in parallel (45s). Pain rating (Numeric Rating Scale 0-10) at 10s, 20s, 30s and 40s of stimulation. The outcome of interest is the a rithmetic mean differences between the Numeric Rating Scale score of the conditioning + test stimulus and test stimulus alone for 4 10s-long epochs (Numeric Rating Scale 0-10) Lower scores indicate better endogenous pain inhibition.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 83 | 82
  Mean change from baseline to 4 months | 0.30 [-0.03 to 0.63] | -0.01 [-0.34 to 0.32]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 69
  Mean change from baseline to 1 year | 0.13 [-0.22 to 0.47] | -0.04 [-0.38 to 0.30]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 80
  Mean change from baseline to 1.5 years | -0.13 [-0.49 to 0.22] | -0.36 [-0.71 to -0.01]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in conditioned pain modulation from baseline to 4 months; Test type: Superiority; p = 0.1948, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.16 to 0.77]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in conditioned pain modulation from baseline to 1 year; Test type: Superiority; p = 0.4937, Multivariate linear model; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.31 to 0.65]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in conditioned pain modulation from baseline to 1.5 years; Test type: Superiority; p = 0.3690, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.27 to 0.73]

9. Secondary Outcome: Self-reported Upper Limb Function
Description: Measured with Disability of Arm, Shoulder and Hand Questionnaire (0-100) with lower scores indicating less disability.
Time Frame: as for outcome 3
Population: Available data differed per timepoints
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 79 | 86
  Mean change from baseline to 4 months | 10.05 [7.05 to 13.05] | 7.81 [4.89 to 10.72]
  Mean change from baseline to 1 year: number analyzed (Participants) | 81 | 83
  Mean change from baseline to 1 year | 8.51 [5.39 to 11.64] | 10.15 [7.07 to 13.22]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 79 | 82
  Mean change from baseline to 1.5 years | 6.56 [3.15 to 9.97] | 9.72 [6.37 to 13.07]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported upper limb function from baseline to 4 months; Test type: Superiority; p = 0.2915, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.24, 95% CI 2-sided [-1.94 to 6.43]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported upper limb function from baseline to 1 year; Test type: Superiority; p = 0.4632, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.63, 95% CI 2-sided [-6.02 to 2.75]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported upper limb function from baseline to 1,5 years; Test type: Superiority; p = 0.1944, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.16, 95% CI 2-sided [-7.94 to 1.63]

10. Secondary Outcome: General Physical Activity Level
Description: Step count average (steps/day) measured with an accelerometer
Time Frame: Postoperatively after 4 months of intensive treatment, at 1 year (after maintenance treatment)
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: steps/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
steps/day
  Mean change from baseline to 4 months: number analyzed (Participants) | 72 | 71
  Mean change from baseline to 4 months | 50 [-600 to 700] | 342 [-316 to 1000]
  Mean change from baseline to 1 year: number analyzed (Participants) | 48 | 48
  Mean change from baseline to 1 year | 1100 [349 to 1850] | 261 [-489 to 1010]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in step count from baseline to 4 months; Test type: Superiority; p = 0.5332, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -293, 95% CI 2-sided [-1218 to 632]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in step count from baseline to 1 year; Test type: Superiority; p = 0.1201, Multivariate linear model; Mean Difference (Net) = 839, 95% CI 2-sided [-221 to 1900]

11. Secondary Outcome: Self-reported Emotional Functioning: Pain Catastrophizing
Description: Measured with the Pain Catastrophizing scale (0-52), with higher scores corresponding to more pain-related catastrophizing.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Geometric Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 79 | 86
  Mean change from baseline to 4 months | 0.896 [0.676 to 1.188] | 1.077 [0.818 to 1.419]
  Mean change from baseline to 1 year: number analyzed (Participants) | 81 | 83
  Mean change from baseline to 1 year | 0.894 [0.679 to 1.176] | 1.065 [0.811 to 1.399]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 80 | 81
  Mean change from baseline to 1.5 years | 0.762 [0.562 to 1.033] | 0.898 [0.663 to 1.216]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain catastrophizing from baseline to 4 months; Test type: Superiority; p = 0.3590, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.831, 95% CI 2-sided [0.561 to 1.233]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain catastrophizing from baseline to 1 year; Test type: Superiority; p = 0.3744, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.839, 95% CI 2-sided [0.570 to 1.236]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported pain catastrophizing from baseline to 1.5 years; Test type: Superiority; p = 0.4533, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = 0.848, 95% CI 2-sided [0.522 to 1.304]

12. Secondary Outcome: Self-reported Emotional Functioning: Depression
Description: Measured with Depression Anxiety Stress scales 21(0-42) with lower scores indicating less depression.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Geometric Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 79 | 84
  Mean change from baseline to 4 months | 0.802 [0.588 to 1.092] | 0.930 [0.558 to 1.330]
  Mean change from baseline to 1 year: number analyzed (Participants) | 82 | 83
  Mean change from baseline to 1 year | 0.625 [0.459 to 0.851] | 0.774 [0.570 to 1.052]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 80 | 82
  Mean change from baseline to 1.5 years | 0.718 [0.535 to 0.963] | 0.749 [0.560 to 1.003]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported depression from baseline to 4 months; Test type: Superiority; p = 0.5018, MUltivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.862, 95% CI 2-sided [0.558 to 1.330]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported depression from baseline to 1 year; Test type: Superiority; p = 0.3362, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.808, 95% CI 2-sided [0.522 to 1.248]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported depression from baseline to 1.5 years; Test type: Superiority; p = 0.8375, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.958, 95% CI 2-sided [0.633 to 1.449]

13. Secondary Outcome: Self-reported Health-related Quality of Life
Description: Measured with the existential well-being sub scale of the McGill Quality of Life questionnaire (0-10) with higher scores reflecting a better health-related quality of life.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 80 | 86
  Mean change from baseline to 4 months | 0.19 [-0.14 to 0.52] | 0.51 [0.19 to 0.84]
  Mean change from baseline to 1 year: number analyzed (Participants) | 82 | 84
  Mean change from baseline to 1 year | 0.90 [0.52 to 1.27] | 0.71 [0.34 to 1.09]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 79 | 83
  Mean change from baseline to 1.5 years | 1.07 [0.64 to 1.49] | 0.61 [0.20 to 1.03]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported health-related quality of life from baseline to 4 months; Test type: Superiority; p = 0.1745, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.78 to 0.14]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported health-related quality of life from baseline to 1 year; Test type: Superiority; p = 0.5025, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.18, 95% CI 2-sided [-0.35 to 0.71]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported health-related quality of life from baseline to 1,5 years; Test type: Superiority; p = 0.1363, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.45, 95% CI 2-sided [-0.14 to 1.05]

14. Secondary Outcome: Socio-economic Outcomes: Return to Work Rate
Description: Work status at 12 and 18 months postoperatively, i.e. the proportion of women working at 12 and 18 months after surgery, respectively
Time Frame: Postoperatively after 1 year (after maintenance treatment) and at 1,5 years (after follow-up)
Population: One hundred fifteen participants (62.5%) were working at time of diagnosis (IG=58; CG=57); available data differed per time point
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 58 | 57
Participants
  At 1 year | 41 [33 to 48] | 30 [22 to 38]
  At 1.5 years | 47 [39 to 53] | 41 [32 to 48]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in proportion of working participants at 1 year; Test type: Superiority; p = 0.074, Fisher Exact; Percentage = -0.184, 95% CI 2-sided [-0.358 to 0.008]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in proportion of working participants at 1,5 years; Test type: Superiority; p = 0.352, Fisher Exact; Percentage = -0.09, 95% CI 2-sided [-0.26 to 0.078]

15. Secondary Outcome: Altered Somatosensory Functions (Temperature-cold)
Description: Thermal detection sensitivity (degrees Celsius) for cold at the arm at the affected side measured with computerized thermotests. Temperature when a change from a thermoneutral state to a distinct cold is recorded.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: degrees Celsius
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
degrees Celsius
  Mean change from baseline to 4 months: number analyzed (Participants) | 83 | 82
  Mean change from baseline to 4 months | -4.77 [-6.47 to -3.08] | -5.00 [-6.70 to -3.31]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 69
  Mean change from baseline to 1 year | -3.36 [-5.00 to -1.71] | -4.16 [-5.81 to -2.52]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 80
  Mean change from baseline to 1.5 years | -3.90 [-5.45 to -2.36] | -4.35 [-5.87 to -2.84]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in cold detection sensitivity from baseline to 4 months; Test type: Superiority; p = 0.8497, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.23, 95% CI 2-sided [-2.17 to 2.64]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in cold detection sensitivity from baseline to 1 year; Test type: Superiority; p = 0.4971, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.81, 95% CI 2-sided [-1.52 to 3.14]
Statistical Analysis 3: Comparison: Intervention Group; Difference in change in cold detection sensitivity from baseline to 1.5 years; Test type: Superiority; p = 0.6831, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.45, 95% CI 2-sided [-1.72 to 2.62]

16. Secondary Outcome: Altered Somatosensory Functions (Nociception: Pinprick Sensation)
Description: Mechanical pain sensitivity (mN) measured at the arm at the affected side with Von Frey Monofilaments. A series of stimulus intensities are given and the stimulus intensity that is first identified as painful (not unbearable) is recorded (mN). Min-max 8mN-512mN.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: mN
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
mN
  Mean change from baseline to 4 months: number analyzed (Participants) | 83 | 82
  Mean change from baseline to 4 months | 19.77 [-17.31 to 56.85] | 14.99 [-22.08 to 52.05]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 69
  Mean change from baseline to 1 year | -22.24 [-59.94 to 15.45] | 35.02 [-2.66 to 72.69]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 79
  Mean change from baseline to 1.5 years | -17.91 [-58.13 to 22.48] | 2.19 [-37.45 to 41.83]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in mechanical pain sensitivity at the arm from baseline to 4 months; Test type: Superiority; p = 0.8584, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 4.78, 95% CI 2-sided [-47.72 to 57.28]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in mechanical pain sensitivity at the arm from baseline to 1 year; Test type: Superiority; p = 0.0353, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -57.25, 95% CI 2-sided [-110.57 to -3.93]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in mechanical pain sensitivity at the arm from baseline to 1.5 years; Test type: Superiority; p = 0.4865, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -20.10, 95% CI 2-sided [-76.72 to 36.52]

17. Secondary Outcome: Altered Somatosensory Functions (Nociception: Deep Pain Sensitivity)
Description: Pressure pain sensitivity (kgf) at the pectoralis region at the affected side measured with an algometer. The amount of pressure (kgs) by which the perception of pressure turns for the first time into a painful (not unbearable) sensation. Lower values indicate higher pain sensitivity.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Mean (95% Confidence Interval); unit: kgf
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
kgf
  Mean change from baseline to 4 months: number analyzed (Participants) | 82 | 82
  Mean change from baseline to 4 months | 1.05 [0.95 to 1.15] | 0.94 [0.86 to 1.03]
  Mean change from baseline to 1 year: number analyzed (Participants) | 70 | 69
  Mean change from baseline to 1 year | 0.84 [0.75 to 0.94] | 0.75 [0.67 to 0.84]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 74 | 80
  Mean change from baseline to 1.5 years | 0.81 [0.73 to 0.91] | 0.78 [0.69 to 0.87]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in pressure pain sensitivity at the pectoral region from baseline to 4 months; Test type: Superiority; p = 0.1278, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.11, 95% CI 2-sided [0.97 to 1.27]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in pressure pain sensitivity at the pectoral region from baseline to 1 year; Test type: Superiority; p = 0.1875, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.11, 95% CI 2-sided [0.95 to 1.30]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in pressure pain sensitivity at the pectoral region from baseline to 1.5 years; Test type: Superiority; p = 0.5612, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.05, 95% CI 2-sided [0.89 to 1.23]

18. Secondary Outcome: Self-reported Emotional Functioning: Anxiety
Description: Measured with Depression Anxiety Stress scales 21 (0-42). Lower scores indicate less anxiety.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Geometric Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 79 | 84
  Mean change from baseline to 4 months | 1.045 [0.772 to 1.415] | 0.987 [0.733 to 1.328]
  Mean change from baseline to 1 year: number analyzed (Participants) | 82 | 83
  Mean change from baseline to 1 year | 0.783 [0.575 to 1.067] | 0.839 [0.617 to 1.138]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 80 | 82
  Mean change from baseline to 1.5 years | 0.829 [0.325 to 1.100] | 0.821 [0.621 to 1.085]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported anxiety from baseline to 4 months; Test type: Superiority; p = 0.7902, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.089, 95% CI 2-sided [0.693 to 1.620]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported anxiety from baseline to 1 year; Test type: Superiority; p = 0.7578, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.934, 95% CI 2-sided [0.604 to 1.443]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported anxiety from baseline to 1.5 years; Test type: Superiority; p = 0.9600, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.010, 95% CI 2-sided [0.679 to 1.504]

19. Secondary Outcome: Self-reported Emotional Functioning: Stress
Description: Measured with Depression Anxiety Stress scales 21 (0-42). Lower scores indicate less stress.
Time Frame: as for outcome 3
Population: Available data differed per time point
Measure: Geometric Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 92 | 92
score on a scale
  Mean change from baseline to 4 months: number analyzed (Participants) | 80 | 84
  Mean change from baseline to 4 months | 0.812 [0.598 to 1.101] | 0.760 [0.563 to 1.026]
  Mean change from baseline to 1 year: number analyzed (Participants) | 82 | 84
  Mean change from baseline to 1 year | 0.782 [0.574 to 1.064] | 0.721 [0.532 to 0.979]
  Mean change from baseline to 1.5 years: number analyzed (Participants) | 80 | 82
  Mean change from baseline to 1.5 years | 0.857 [0.629 to 1.167] | 0.868 [0.639 to 1.178]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in change in self-reported stress from baseline to 4 months; Test type: Superiority; p = 0.7619, Multivariate linear model; multivariate linear model for longitudinal measures with an unstructured covariance matrix was applied for each continuous outcome; Mean Difference (Net) = 1.068, 95% CI 2-sided [0.696 to 1.639]
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Difference in change in self-reported stress from baseline to 1 year; Test type: Superiority; p = 0.7169, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.087, 95% CI 2-sided [0.702 to 1.673]
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Difference in change in self-reported stress from baseline to 1.5 years; Test type: Superiority; p = 0.9535, Multivariate linear model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.987, 95% CI 2-sided [0.639 to 1.525]

ADVERSE EVENTS:
Time Frame: Total study duration, i.e. 1.5 years
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/92 | 1/92
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/92 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03351075/Prot_SAP_000.pdf